CLINICAL TRIAL: NCT02224105
Title: Safety, Tolerability, Pharmacodynamics and Pharmacokinetics of a BI 653048 BS H3PO4 Capsule Formulation Administered as Multiple Doses of 25 mg to 200 mg Once Daily (qd) for 3 Days Assessing Pharmacodynamics as Endotoxin-induced Inflammatory Response of a Single Intravenous Bolus Administration of 2 ng/kg Body Weight Lipopolysaccharide (LPS). A Randomised, Double-blind Within Dose Groups, Placebo-controlled, Multiple Rising Dose Phase I Trial With Open-label Active Comparator in Healthy Male Subjects
Brief Title: Safety, Tolerability, Pharmacodynamics and Pharmacokinetics of BI 653048 BS H3PO4 Capsule Assessing Endotoxin-induced Inflammatory Response in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1262.9
Record Dates: First submitted 2014-08-21; First posted 2014-08-25 (Estimated); Last update posted 2014-08-25 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
MeSH Terms: interventions — BI 653048 BS H3PO4; endotoxin, Escherichia coli; Lipopolysaccharides

ARMS (4):
- BI 653048 BS (Experimental): escalating doses
  Interventions: Drug: BI 653048 BS; Drug: sodium chloride infusion; Drug: endotoxin escherichia coli (E. coli) lipopolysaccharide (LPS)
- Prednisolone low (Active Comparator)
  Interventions: Drug: Prednisolone low; Drug: sodium chloride infusion; Drug: endotoxin escherichia coli (E. coli) lipopolysaccharide (LPS)
- Prednisolone high (Active Comparator)
  Interventions: Drug: Prednisolone high; Drug: sodium chloride infusion; Drug: endotoxin escherichia coli (E. coli) lipopolysaccharide (LPS)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: sodium chloride infusion; Drug: endotoxin escherichia coli (E. coli) lipopolysaccharide (LPS)

INTERVENTIONS:
Drug: BI 653048 BS
  Arms: BI 653048 BS
Drug: Prednisolone low
  Arms: Prednisolone low
Drug: Prednisolone high
  Arms: Prednisolone high
Drug: Placebo
  Arms: Placebo
Drug: sodium chloride infusion
Drug: endotoxin escherichia coli (E. coli) lipopolysaccharide (LPS)

SUMMARY:
The general aim of the current study was to investigate the safety and tolerability, and pharmacodynamics (endotoxin-induced inflammatory response of a single intravenous bolus administration of 2 ng/kg body weight Escherichia coli lipopolysaccharide (LPS)) of BI 653048 BS H3PO4 capsules in healthy male subjects following oral administration of multiple rising doses of 25 mg to 200 mg over three days compared to the active comparator prednisolone and placebo.

Pharmacodynamics were assessed by investigating the influence of LPS administration on inflammatory parameters. More specifically, it was evaluated whether and to what extent the symptoms induced by LPS challenge can be attenuated by ascending BI 653048 BS H3PO4 doses using prednisolone as positive control and placebo as negative control. A secondary objective was the exploration of pharmacokinetics of BI 653048 BS, the investigation of other pharmacodynamic parameters (biomarker) and of the tolerability of LPS.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males according to the following criteria:

   Based upon a complete medical history, including the physical examination, vital signs (blood pressure, pulse rate and body temperature), 12-lead ECG, clinical laboratory tests
2. Age ≥18 and Age ≤50 years
3. Body mass index (BMI) ≥18.5 and BMI ≤29.9 kg/m2
4. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local legislation

Exclusion Criteria:

1. Any finding of the medical examination (including blood pressure, pulse rate, orthostatic test, body temperature and ECG) deviating from normal and of clinical relevance
2. Any evidence of a clinically relevant concomitant disease
3. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
4. Surgery of the gastrointestinal tract (except appendectomy)
5. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
6. History of relevant orthostatic hypotension, fainting spells or blackouts
7. Chronic or relevant acute infections
8. History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
9. Intake of drugs with a long half-life (>24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
10. Use of drugs which might reasonably influence the results of the trial or that prolong the QT/QTc interval based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
11. Participation in another trial with an investigational drug within 30 days prior to administration or during the trial
12. Smoker (>10 cigarettes or >3 cigars or >3 pipes/day)
13. Inability to refrain from smoking for 1 day prior to first drug administration until discharge from the study site
14. Alcohol abuse (more than 60 g/day)
15. Drug abuse
16. Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
17. Excessive physical activities (within one week prior to administration or during the trial)
18. Any laboratory value outside the reference range that is of clinical relevance
19. Inability to comply with dietary regimen of trial site

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2010-03; Primary Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events | up to 37 days
Number of subjects with clinically significant findings in vital signs | up to day 15
  blood pressure, pulse rate and body temperature
Number of subjects with clinically significant findings in 12-lead electrocardiogram (ECG) | up to day 15
Number of subjects with clinically significant findings in laboratory tests | up to day 15
Assessment of tolerability by investigator on a 4-point scale | up to day 15
Maximum measured concentration of the biomarker level in plasma (Emax) | up to 96 hours after first drug administration
Area under the concentration-time curve of the biomarker in plasma over the time interval from 0 to the last measurable time point of the dose (AUEC) | up to 96 hours after first drug administration

SECONDARY OUTCOMES:
Maximum measured concentration of the analyte in plasma at steady state (Cmax,ss) | up to 96 hours after first drug administration
Time from dosing to maximum measured concentration of the analyte at steady state (tmax,ss) | up to 96 hours after first drug administration
Area under the concentration-time curve of the analyte in the plasma over the time interval from 0 to the last measurable time point of the dose at steady state (AUC0-tz,ss) | up to 96 hours after first drug administration
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity at steady state (AUC0-∞,ss) | up to 96 hours after first drug administration
Percentage of the AUC0-∞ that is obtained by extrapolation at steady state (%AUCtz-∞,ss) | up to 96 hours after first drug administration
Terminal phase elimination rate constant at steady state (λz,ss) | up to 96 hours after first drug administration
Terminal phase elimination half life at steady state (t1/2,ss) | up to 96 hours after first drug administration
Mean residence time of the analyte in the body after oral administration at steady state (MRTpo,ss) | up to 96 hours after first drug administration
Apparent clearance of the analyte in plasma following extravascular administration at steady state (CL/Fss) | up to 96 hours after first drug administration
Apparent volume of distribution during the terminal phase λz following an extravascular dose at steady state (Vz/Fss) | up to 96 hours after first drug administration
Minimum measured concentration of the biomarker during the treatment interval (Emin) | up to 96 hours after first drug administration
Area under the concentration-time curve of the biomarker in serum over the time interval from 0 to the last measurable time point of the dose (AUEC) | up to 96 hours after first drug administration
Measured concentration of the biomarker at time t after the beginning of the treatment interval (Et) | up to 96 hours after first drug administration

REFERENCES:
- [Derived] Harcken C, Scholl P, Nabozny G, Thomson D, Bianchi D. Clinical profile of the functionally selective glucocorticoid receptor agonist BI 653048 in healthy male subjects. Expert Opin Investig Drugs. 2019 May;28(5):489-496. doi: 10.1080/13543784.2019.1599859. Epub 2019 Apr 9. PMID 30908082